CLINICAL TRIAL: NCT03132298
Title: Effects of a Single-session Implicit Theories of Personality Intervention on Recovery From Social Stress and Long-term Psychological Functioning in Early Adolescents
Brief Title: Effects of a Single-session Implicit Theories of Personality Intervention on Early Adolescent Psychopathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); American Psychological Foundation (Other)
Responsible Party: Principal Investigator, Jessica Schleider, PhD candidate, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB15-0855; 1F31MH108280-01 (NIH); 5F31MH108280-02 (NIH)
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Results first posted 2019-01-23 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-01

CONDITIONS: Anxiety Symptoms; Depressive Symptoms
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Participants (N=96), ages 12-15 will be randomized to receive one of two a 30-minute, computer-based programs: (1) a 'growth mindset' program, teaching that personal traits and characteristics are malleable; or (2) a control program, designed to mimic 'supportive therapy,' teaching the value of sharing one's feelings with close others.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implicit Theories of Personality Program (Experimental): This program is self-administered, computer-based, and 30 minutes in length. Content is designed to maximize relevance for youths with internalizing distress. The program includes 5 elements: 1. An introduction the concept of neuroplasticity; 2. Testimonials from older youths describing beliefs that people's traits are malleable, given the brain's capacity for change; 3. Further vignettes by older youths describing times when they used "growth mindsets" to cope with peer rejection, hopelessness, and feared embarrassment; 4. A worksheet describing strategies for applying these principles to participants' lives; 5. An exercise wherein participants write notes to younger children, using newly-gleaned information about the malleability of personal traits to help them to cope with setbacks
  Interventions: Other: Implicit Theories of Personality Program
- Control Program (Active Comparator): The Control Program is a computer-based session of supportive therapy (ST), designed to encourage youths to identify and express feelings. ST does not teach specific skills or beliefs and has been shown to be less effective than cognitive-behavioral interventions in reducing youth internalizing distress. Here, ST was designed to control for nonspecific intervention elements (eg. completing an interactive computer program) and to encourage youths to share emotions with others. ST included the same number of reading/writing activities as the experimental program and took the same amount of time (30 mins.) to complete.
  Interventions: Other: Control Program

INTERVENTIONS:
Other: Implicit Theories of Personality Program — This 30-minute, self-administered computer program teaches youths that personality is malleable, as opposed to fixed, due to the human brain's constant potential for change and growth (i.e., neuroplasticity).
  Other Names: Growth Mindset of Personality Program
  Arms: Implicit Theories of Personality Program
Other: Control Program — This 30-minute, self-administered computer program was designed to control for nonspecific aspects of completing a series of computer-based activities in the context of the present study. It was also designed to mimic 'supportive therapy' that youths might receive in usual care settings, stressing the importance of sharing one's feelings with close others.
  Other Names: Supportive Therapy (ST) Program
  Arms: Control Program

SUMMARY:
The goal of the project is to test whether a single-session intervention teaching incremental theories of personality, or the belief that one's personality is malleable, can strengthen recovery from social stress and reduce the development of anxiety and depression during early adolescence. Results may suggest a scalable, cost-effective approach to improving youths' coping capacities and preventing adverse mental health outcomes over time.

DETAILED DESCRIPTION:
Efforts to prevent and reduce mental health problems in youths have advanced greatly in recent years. However, these advances have not reduced rates of youth mental illness on a large scale. Thus, a great need exists for novel, scalable, and low-cost approaches to reducing mental health problems in youth. Ideally, such approaches would be mechanism-targeted: that is, they would act on specific developmental processes that underlie psychological disorders. The proposed research aims to address this need by testing whether a single-session intervention teaching incremental theories of personality, or the belief that one's personality is malleable-as opposed to entity theories of personality, or the belief that one's personality is fixed and unchangeable-can strengthen recovery from social stress and prevent the development of anxiety and depression during early adolescence. Compared to incremental theories, entity theories of personal traits have demonstrated cross-sectional and prospective relations with greater anxiety and depression in youths. Further, a single-session incremental personality theories intervention reduced the development of depressive symptoms in a community sample of adolescents, supporting these theories as powerful intervention and/or prevention targets, even when taught in a brief format. Specifically, this project has two aims. Aim 1 is to evaluate the effect of the implicit theories intervention on two candidate mechanisms of action, or targets, identified by prior research: arousal (measured via physiological reactivity following social stress) and loss (here, perceived loss of behavioral control) in youths 12-15 years of age. Following a lab-based social stress induction, I hypothesize that participants receiving the intervention will recover from stress more rapidly, as indicated by measures of arousal (heart rate variability; electrodermal activity levels) and self-reported loss (increased self-reported perceived control) compared to participants who do not receive the intervention. Aim 2 is to evaluate the effects of the single-session incremental theories intervention on anxiety and depression over a nine-month follow-up period. I will test whether the intervention, compared to a control protocol, reduces symptoms of anxiety an depression the development of anxiety and depression; I will also assess whether this change is a direct result of shifts in the two aforementioned targets (arousal; loss). I predict more positive trajectories in anxiety and depression for youth receiving the intervention, relative to those who do not receive the intervention, across nine months. I will also test whether these trajectories are mediated by changes in the targets described in Aim 1. Finally, regardless of outcomes for Aims 1 and 2, baseline, postintervention, and 9-month measures will be used to map links among implicit theories, interventions targeting those theories, social stress recovery, and youth anxiety and depression over time. Findings may suggest a cost-effective, scalable intervention that improves youth resiliency and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12 to 15 (inclusive) at time of study enrollment
* One or more of the following (3) criteria, all assessed through an initial parent phone screen: (1) t-score of >60 (84th percentile) on any disorder subscale of the Revised Child Anxiety and Depression Scale-Parent (RCADS-P, Ebesutani et al., 2010); (2) school-based accommodations for anxiety- or depression-related symptoms, such as through an Individual Education Plan (IEP) or a 504 plan; (3) anxiety and/or depression treatment sought for the youth within the previous 3 years.

Exclusion Criteria:

* Psychosis, intellectual disability, pervasive developmental/autism spectrum disorder, and suicidal ideation leading to hospitalization or attempts within the past year.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Schleider, M.A., Principal Investigator — Harvard University
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing plan is consistent with NIH guidelines for sharing participant-level data at the conclusion of the fellowship period.

REFERENCES:
- [Result] Schleider JL, Weisz JR. Reducing risk for anxiety and depression in adolescents: Effects of a single-session intervention teaching that personality can change. Behav Res Ther. 2016 Dec;87:170-181. doi: 10.1016/j.brat.2016.09.011. Epub 2016 Sep 26. PMID 27697671
- [Derived] Schleider JL, Abel MR, Weisz JR. Do Immediate Gains Predict Long-Term Symptom Change? Findings from a Randomized Trial of a Single-Session Intervention for Youth Anxiety and Depression. Child Psychiatry Hum Dev. 2019 Oct;50(5):868-881. doi: 10.1007/s10578-019-00889-2. PMID 30993499
- [Derived] Schleider J, Weisz J. A single-session growth mindset intervention for adolescent anxiety and depression: 9-month outcomes of a randomized trial. J Child Psychol Psychiatry. 2018 Feb;59(2):160-170. doi: 10.1111/jcpp.12811. Epub 2017 Sep 18. PMID 28921523

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implicit Theories of Personality Program | Control Program
Started | 48 | 48
Completed | 36 | 35
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Implicit Theories of Personality Program | Control Program | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 48 | 96
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.39 (1.58) | 13.26 (1.06) | 13.33 (1.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 22 | 21 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 48 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Children's Depression Inventory (CDI) From Baseline to 9-month Follow-up
Description: the Children's Depression Inventory, a 27-item self-report questionnaire that measures cognitive, affective, and behavioral symptoms of depression. Items are scored from 0-2, and scores range from 0 to 44; higher scores indicate greater symptom severity. The CDI is reliable and valid. It can distinguish youths with more or less severe depressive symptoms, as well as youths at risk for depression from non-depressed youths. Suicide- and self-harm related questions were removed for the purposes of this study.
Time Frame: Baseline and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
scores on a scale
  Baseline CDI-C scores | 12.35 (1.05) | 11.76 (1.07)
  3-month CDI-C scores | 11.54 (1.07) | 11.66 (1.14)
  6-month CDI-C scores | 10.85 (1.16) | 12.74 (1.21)
  9-month CDI-C scores | 10.19 (1.36) | 12.47 (1.39)

2. Primary Outcome: Change in Children's Depression Inventory - Parent (CDI-P) From Baseline to 9-month Follow-up
Description: the Children's Depression Inventory, a 27-item self-report questionnaire that measures cognitive, affective, and behavioral symptoms of depression. Items are scored from 0-2, and scores range from 0 to 44; higher scores indicate greater symptom severity. The CDI and the parent analog (CDI-P) is reliable and valid. It can distinguish youths with more or less severe depressive symptoms, as well as youths at risk for depression from non-depressed youths. Suicide- and self-harm related questions were removed for the purposes of this study.
Time Frame: Baseline and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
scores on a scale
  Baseline CDI-P scores | 13.53 (1.05) | 11.27 (0.96)
  3-month CDI-P scores | 11.41 (0.97) | 10.19 (0.95)
  6-month CDI-P scores | 10.61 (0.94) | 9.51 (0.94)
  9-month CDI-P scores | 9.69 (0.87) | 10.84 (1.01)

3. Primary Outcome: Change in Screen for Child Anxiety Related Disorders - Child (SCARED-C) From Baseline to 9-month Follow-up
Description: Anxiety symptoms were assessed at baseline and at each follow-up point using the Screen for Child Anxiety and Related Disorders - Child and Parent versions (SCARED-C/SCARED-P). The SCARED-C and SCARED-P are child and parent versions of the same 41-item questionnaire measure of pediatric anxiety. Both differentiate between clinically anxious and nonanxious psychiatrically ill youth. Youths/parents respond to items using a 3-point Likert scale describing the degree to which statements are true about them; scores range from 0 to 82. Internal consistency, test-retest reliability, and construct validity of the SCARED are strong (Hale, Raaijmakers, Muris, & Meeus, 2005; Myers & Winters, 2002). In this study, the SCARED-C/P Total Scores were used and derived by summing all 41 items, with higher scores reflecting higher levels of anxiety.
Time Frame: Baseline and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
score on a scale
  Baseline SCARED-C scores | 28.13 (2.05) | 30.54 (2.10)
  3-month SCARED-C scores | 24.43 (2.21) | 30.47 (2.34)
  6-month SCARED-C scores | 24.25 (2.23) | 29.76 (2.33)
  9-month SCARED-C scores | 23.12 (2.43) | 30.44 (2.49)

4. Primary Outcome: Change in Screen for Child Anxiety Related Disorders - Parent (SCARED-P) From Baseline to 9-month Follow-up
Description: Anxiety symptoms were assessed at baseline and at each follow-up point using the Screen for Child Anxiety and Related Disorders - Child and Parent versions (SCARED-C/SCARED-P). The SCARED-C and SCARED-P are child and parent versions of the same 41-item questionnaire measure of pediatric anxiety. Both differentiate between clinically anxious and nonanxious psychiatrically ill youth. Youths/parents respond to items using a 3-point Likert scale describing the degree to which statements are true about them; scores range from 0 to 82. Internal consistency, test-retest reliability, and construct validity of the SCARED are strong. In this study, the SCARED-C/P Total Scores were used and derived by summing all 41 items, with higher scores reflecting higher levels of anxiety.
Time Frame: Baseline and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
score on a scale
  Baseline SCARED-P scores | 25.56 (1.42) | 25.24 (1.48)
  3-month SCARED-P scores | 22.31 (1.38) | 21.65 (1.74)
  6-month SCARED-P scores | 16.65 (1.27) | 18.23 (1.70)
  9-month SCARED-P scores | 18.07 (1.74) | 20.99 (1.93)

5. Secondary Outcome: Primary Control Scale for Children (PCSC)
Description: The PCSC is a 24-item scale measuring perceived ability to exert primary control: to influence or alter objective events or conditions through personal effort. Participants rated agreement with statements about their ability to exert primary control, with half the items worded in a positive direction (e.g., "I can do well on tests if I study hard.") and half in a negative direction (e.g., "I cannot get other kids to like me no matter how hard I try."). Responses range from "very true" to "very false" on a four-point Likert scale. Scores range from 0 to 72, with higher scores indicating higher (more adaptive) levels of perceived primary control.
Time Frame: Baseline, immediately post-intervention, and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
score on a scale
  Baseline PCSC | 55.60 (1.43) | 56.17 (1.46)
  Immediate Post-Intervention PCSC | 59.17 (1.40) | 56.07 (1.42)
  3-month PCSC | 59.49 (1.42) | 55.89 (1.58)
  6-month PCSC | 57.50 (1.59) | 56.56 (1.69)
  9-month PCSC | 58.81 (1.64) | 55.04 (1.65)

6. Secondary Outcome: Secondary Control Scale for Children (SCSC)
Description: The SCSC is a 20-item scale measuring perceived ability to exert secondary control: to influence the personal psychological impact of objective conditions on oneself, by adjusting oneself to fit those conditions. Item content reflects response patterns associated with various kinds of secondary control, such as finding a silver lining ("I can usually find something good to like, even in a bad situation.") and adjusting cognition ("When something bad happens, I can find a way to think about it that makes me feel better."). Respondents rate agreement with each item on a 4-point Likert scale from "very false" to "very true." Scores range from 0-60, with higher scores corresponding to higher (more adaptive) levels of perceived secondary control.
Time Frame: Baseline, immediately post-intervention, and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
score on a scale
  Baseline SCSC | 33.25 (1.72) | 33.32 (1.75)
  Immediate Post-Intervention SCSC | 36.56 (1.62) | 34.09 (1.42)
  3-month SCSC | 36.99 (1.71) | 32.91 (1.83)
  6-month SCSC | 34.59 (1.79) | 33.14 (1.86)
  9-month SCSC | 34.41 (2.05) | 31.37 (2.09)

7. Secondary Outcome: Electrodermal Activity (EDA) Recovery Slope
Description: EDA was assessed continuously during the laboratory baseline (5 min prior to the social stress induction), social stress induction, and recovery period (5 min following the social stress induction) using Biopac MP150 hardware at a sampling rate of 1000 readings persecond and a 0.5e1 Hz bandpass filter. EDA was measured with a Biopac GSR100C amplifier and two EDA isotonic gel electrodes placed on the thenar and hypothenar eminences of the child's nondominant hand. EDA data were acquired and analyzed using AcqKnowledge 4.1 Software. Research assistants trained by the first author manually identified and removed artifacts. Averages (expressed in micro-Siemens) for EDA during the baseline, speech preparation, speech, and recovery periods were calculated for each participant. Slopes of EDA change during the recovery were calculated, expressed in microSiemens per second.
Time Frame: Assessed at immediate post-intervention only
Measure: Mean (Standard Deviation); unit: microsiemens/second
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 44 | 43
microsiemens/second | -.00082 (0.011) | -.00024 (0.013)

8. Secondary Outcome: Heart Rate Variability (HRV) Recovery Slope
Description: HRV was assessed; specifically, the time-based root-mean square successive difference of normal-to-normal (N-to-N) intervals (rMSSD). RMSSD equates to mean shifts in the time elapsed between consecutive heartbeats, in milliseconds. It reflects parasympathetically mediated, short-term changes in HRV. More rapid post-stressor increases in rMSSD (during the 5-min post stressor recovery period) indicated a more adaptive recovery trajectory following stress. Here, rMSSD was computed using the Acqknowledge automated time-series HRV analysis function.
Time Frame: Assessed at immediate post-intervention only
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 36 | 40
msec | .008 (.034) | -.007 (.040)

9. Other Pre Specified Outcome: Beck Depression Inventory
Description: Parental depressive symptoms were measured at baseline at 3-, 6-, and 9-month follow-up assessments using the Beck Depression Inventory-II (BDI-II). The BDI is one of the most widely used and evaluated self- report measures of adult depressive symptoms. For each of its 21 items, respondents select among four alternative responses reflecting the increasing levels of symptom severity (0 = no symptom present to 3 = severe symptom present). The total score was used in this study, with a possible score range of 0 to 63 at each assessment point. Higher scores indicate higher levels of depressive symptoms.
Time Frame: Baseline and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
score on a scale
  BDI baseline | 7.92 (8.19) | 6.91 (6.26)
  BDI 3-month | 8.61 (9.66) | 10.89 (10.75)
  BDI 6-month | 7.54 (7.38) | 7.80 (9.00)
  BDI 9-month | 6.74 (6.48) | 7.44 (6.82)

10. Other Pre Specified Outcome: Beck Anxiety Inventory
Description: Parental anxiety symptoms were measured at baseline at 3-, 6-, and 9-month follow-up assessments using the Beck Anxiety Inventory (BAI; Beck & Steer, 1993), a widely-used self-report measure of anxiety in adults for use in clinical, community, and research settings. Respondents report the extent to which they have been bothered by each of 21 symptoms over the preceding week. Each item has four possible answer choices: Not at All; Mildly; Moderately, and Severely. Because the BAI's 21 items (each rated 0 to 3, for a total possible scores ranging from 0 to 63 - higher scores indicate higher levels of anxiety) describe the emotional, physiological, and cognitive symptoms of anxiety but not depression, it can discriminate anxiety from depression in adults.
Time Frame: Baseline and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
score on a scale
  BAI Baseline | 8.60 (9.20) | 6.57 (7.20)
  BAI 3 month | 11.48 (9.89) | 9.58 (13.51)
  BAI 6 month | 5.51 (5.64) | 3.68 (3.92)
  BAI 9 month | 6.23 (5.41) | 5.47 (6.75)

11. Other Pre Specified Outcome: Brief Family Assessment Measure
Description: The BFAM is a 14-item parent report questionnaire assessing perceptions of family functioning during the previous 2 weeks. This instrument was created to provide an operational definition and means of measuring the seven constructs in the Process Model of Family Functioning; it includes two items relating to each construct. Items such as "We take the time to listen to each other" and "When things aren't going well it takes too long to work them out" are scored on a 5-point scale. Items are summed to create a total score (range: 0-70), with higher scores indicating greater familial dysfunction.
Time Frame: Baseline and 3-, 6-, and 9-month (final) follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
score on a scale
  BFAM baseline | 10.60 (4.89) | 11.48 (6.95)
  BFAM 3 months | 10.88 (5.11) | 12.86 (5.66)
  BFAM 6 months | 11.38 (6.30) | 13.00 (5.84)
  BFAM 9 months | 10.29 (5.31) | 12.44 (6.94)

12. Other Pre Specified Outcome: Implicit Personality Theory Questionnaire
Description: The Implicit Personality Theory Questionnaire asks participants to indicate on a 1 (really disagree) to 6 (really agree) scale the extent to which they endorse three statements: "You have a certain personality, and it is something that you can't do much about"; "Your personality is something about you that you can't change very much"; and "Either you have a good personality or you don't, and there is really very little you can do about it." Numerical scores are summed to yield a single, total implicit theory of personality score (score range=0-18); higher scores indicate a stronger entity theory of personality, and lower scores indicate stronger incremental theories of personality.
Time Frame: Baseline, immediately post-intervention, and 3-, 6-, and 9-month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implicit Theories of Personality Program | Control Program
Number analyzed (Participants) | 48 | 48
score on a scale
  Implicit Theories basline | 10.98 (3.15) | 9.93 (3.02)
  Implicit Theories post intervention | 6.77 (3.83) | 8.69 (3.25)
  Implicit Theories 3 month follow-up | 9.72 (3.36) | 9.91 (4.16)
  Implicit Theories 6 month follow-up | 8.75 (2.93) | 10.06 (3.51)
  Implicit Theories 9 month follow-up | 9.23 (3.55) | 10.28 (3.78)

ADVERSE EVENTS:
Arm/Group | Implicit Theories of Personality Program | Control Program
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No